CLINICAL TRIAL: NCT04215744
Title: An Observational Study About Nail Changes Associated With Adjuvant/Neo-adjuvant Chemotherapy and a Prospective Phase II Study About Prevention of Chemotherapy-related Nail Pigmentation by Ice Water Immersion in Breast Cancer Patients
Brief Title: Nail Changes Associated With Chemotherapy and Prevention of Nail Pigmentation by Ice Water Immersion
Acronym: NIPPER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xu fei, Associate Chief Physician, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYSU003-2020
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: self-control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ice water immersion group (Experimental): Ice water immersion of the left hands(30 minutes before the infusion, during the infusion, and 30 minutes after the end of infusion).
  Interventions: Behavioral: Ice water immersion
- Control group (No Intervention): No intervention of the right hands as control.

INTERVENTIONS:
Behavioral: Ice water immersion — Ice water immersion of the left hands
  Arms: Ice water immersion group

SUMMARY:
Anthracyclines combined with cyclophosphamide or taxane-containing regimens may cause nail pigmentation which reduces quality of life in breast cancer patients. We conducted this study to investigate nail pigmentation and other skin changes associated with these drugs and aim to evaluate the effect of ice water immersion of hands on nail pigmentation. The first phase is an observational study. Breast cancer patients who received anthracyclines combined with cyclophosphamide or taxane-containing regimens for adjuvant/neoadjuvant chemotherapy are enrolled. The second phase is a prospective phase II study. Early breast cancer patients who plan to receive these drugs for adjuvant/neoadjuvant chemotherapy are treated with ice water immersion of the left hands while their right hands serve as control. The primary end point is the degree of nail pigmentation. The other end points are the incidence of nail pigmentation in both hands, the degree and the incidence of onycholysis, the time from the first chemotherapy to the occurrence of nail pigmentation/onycholysis, the recovery of nail pigmentation/onycholysis, and patient comfort.

DETAILED DESCRIPTION:
Anthracyclines combined with cyclophosphamide or taxane-containing regimens are commonly used for adjuvant or neoadjuvant chemotherapy in breast cancer patients. However, these drugs may cause nail pigmentation which reduces quality of life in patients. We conducted this study to investigate nail pigmentation and other skin changes associated with anthracyclines in combination with cyclophosphamide or taxane-containing regimens in breast cancer patients who received adjuvant or neoadjuvant chemotherapy. Besides, we aim to evaluate the effect of ice water immersion of hands on nail pigmentation caused by chemotherapy.

The first phase is an observational study. Breast cancer patients who received anthracyclines combined with cyclophosphamide or taxane-containing regimens for adjuvant or neoadjuvant chemotherapy were followed up until six months after the last course of chemotherapy. The second phase is a prospective phase II study. Early breast cancer patients who plan to receive anthracyclines combined with cyclophosphamide or taxane-containing regimens for adjuvant or neoadjuvant chemotherapy are treated with ice water immersion of the left hands while their right hands serve as control. The primary end point is the degree of nail pigmentation. The other end points are the incidence of nail pigmentation in both hands, the degree and the incidence of onycholysis, the time from the first chemotherapy to the occurrence of nail pigmentation/onycholysis, the recovery of nail pigmentation/onycholysis, and patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Early breast cancer patients who plan to receive anthracyclines combined with cyclophosphamide or taxane-containing regimens for adjuvant/neoadjuvant chemotherapy
* No previous nail or skin abnormalities
* No upper limb defects
* Have not received any antitumor treatments before

Exclusion Criteria:

* Have any mental condition that prevents the understanding of the contents of this study and can't complete the study or provide the information required.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Degree of nail pigmentation | 1 year
  Score according to the area of the nail bed where the pigmentation occurs and the color depth:
  Area score: 0 (no change), 1 (1/3 area of nail bed), 2 (2/3 area), 3 (3/3 area); Color score: 0 (no change), 1 (light), 2 (gray), 3 (black). The most severe finger is selected to score.

SECONDARY OUTCOMES:
Degree of onycholysis | 1 year
  According to National Cancer Institute Common Toxicity Criteria; that is, grade 1, indicated by discoloration, ridging (koilonychia), or pitting; and grade 2, indicated by partial or complete onycholysis or pain in the nail bed.
Incidence of nail pigmentation | 1 year
  As long as one finger has nail pigmentation, it is regarded that one patient has nail pigmentation.
Incidence of onycholysis | 1 year
  As long as one finger has onycholysis, it is regarded that one patient has onycholysis.

OTHER OUTCOMES:
Patient comfort | 1 year
  Patients' comfort level is assessed using a 4-point rating system that determined whether patients were dissatisfied (0), not very satisfied (1), satisfied (2), or very satisfied (3)
Occurrence time of nail pigmentation/onycholysis | 1 year
  Defined as the time from the first chemotherapy to the occurrence of nail pigmentation/onycholysis.
Recovery time of nail pigmentation/onycholysis | 1 year
  Defined as the time from the occurrence to the recovery of nail pigmentation/onycholysis.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Xu, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No